CLINICAL TRIAL: NCT00207753
Title: Efficacy and Nutritional Assessment Following Albendazole and Combined Albendazole/Ivermectin Treatment for Intestinal Helminth Infections in Rural Guatemalan Schoolchildren
Brief Title: Effectiveness of Combined Albendazole and Ivermectin Treatment for Intestinal Worm Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Universidad del Valle, Guatemala (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-NCID-4283
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-11-17 (Estimated); Status verified 2005-09

CONDITIONS: Ascariasis; Trichuriasis; Hookworm Infection; Strongyloidiasis; Pediculosis
Keywords: ascaris; trichuris; strongyloides; hookworm; head lice
MeSH Terms: conditions — Ascariasis; Trichuriasis; Hookworm Infections; Strongyloidiasis; Lice Infestations; Ancylostomiasis

INTERVENTIONS:
Drug: albendazole vs. combined albendazole/ivermectin treatment

SUMMARY:
The aim of this study is to compare the efficacy and impact on growth of two drug treatments against intestinal worms in schoolchildren from a rural area of Guatemala. According to the World Bank, these intestinal worms are one of the top causes of childhood health problems in many areas of the developing world (The World Bank, 1993). Infected children are more likely to have inadequate nutrition due to the worm infections and are more likely to be shorter in height and weigh less than children who are not infected. After collecting height and weight information, we will split the children into two groups. One group will receive albendazole and the other group will receive combined albendazole/ivermectin. Both groups will be receiving albendazole, the current standard of care treatment. Ivermection is expected to improve efficacy and nutritional benefit as well as add increased scope of treatment for the worm Strongyloides, and ectoparasites such as scabies and head lice. Both treatment regimens and the combination have been used millions of times in the developing world and are safe to use. Co-administration of drugs would be a more efficient use of the opportunity to access schoolchildren and provide deworming treatment.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy and nutritional impact of two drug treatments against intestinal helminths from a rural area of Guatemala. The helminths that will be analyzed in this study are Ascaris lumbricoides, Trichuris trichiura, and hookworm. Because of the manifestations of these helminths infections, nutritional status can deteriorate in infected persons. According to the World Bank, these helminths are one of the top causes of childhood morbidity in many areas of the developing world (The World Bank, 1993).

This information will be gathered by collecting stool samples from schoolchildren, in order to determine the prevalence of infection in children living around Poptun, Guatemala. Height and weight measurements will also be taken, along with a visual exam of the skin for other parasitic skin infections. Children with an inadequate nutritional status are likely to be shorter in height and weigh less than children reared in an area with a low prevalence of helminths. After collecting this baseline information, we will split the children into two groups. One group will receive albendazole and the other group will receive albendazole/ivermectin. Both groups will be receiving is albendazole, the current standard of care treatment. Ivermectin is expected to improve efficacy and nutritional benefit as well as adding increased scope of treatment (Strongyloides, ectoparasites such as scabies and head lice). Both treatment regimens and the combination have been used millions of times in the developing world and are safe to use. Co-administration of drugs is thought to be a more efficient use of the opportunity to access schoolchildren and provide health improvements. Providing data to support expanded treatment options will provide public health officials with the data needed to make such decisions.

ELIGIBILITY:
Inclusion Criteria:

Children will be eligible to participate in the study if they are between 5 and 12 years of age, are students in schools selected for study, and if parental consent and child assent for participation has been obtained.

Exclusion Criteria:

those not fitting criteria above

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 550
Dates: Start 2005-02; Study Completion 2005-03

PRIMARY OUTCOMES:
efficacy against geohelminths (stool egg count)
height increase
weight increase

SECONDARY OUTCOMES:
ectoparasite examination

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Beach, Ph.D., Principal Investigator — Centers for Disease Control and Prevention; Byron Arana, MD, Principal Investigator — MERTU/CDC-Universite de Valle de Guatemala
Locations (1):
- Various elementary schools, Poptún, Departamento del Petén, Guatemala

REFERENCES:
- [Background] Stephenson LS, Latham MC, Ottesen EA. Global malnutrition. Parasitology. 2000;121 Suppl:S5-22. doi: 10.1017/s0031182000006478. PMID 11386691
- [Background] Stephenson LS, Latham MC, Ottesen EA. Malnutrition and parasitic helminth infections. Parasitology. 2000;121 Suppl:S23-38. doi: 10.1017/s0031182000006491. PMID 11386688
- [Background] Horton J, Witt C, Ottesen EA, Lazdins JK, Addiss DG, Awadzi K, Beach MJ, Belizario VY, Dunyo SK, Espinel M, Gyapong JO, Hossain M, Ismail MM, Jayakody RL, Lammie PJ, Makunde W, Richard-Lenoble D, Selve B, Shenoy RK, Simonsen PE, Wamae CN, Weerasooriya MV. An analysis of the safety of the single dose, two drug regimens used in programmes to eliminate lymphatic filariasis. Parasitology. 2000;121 Suppl:S147-60. doi: 10.1017/s0031182000007423. PMID 11386686
- [Background] World Health Organization, 1992. Health of school children: treatment of intestinal helminths and schistosomiasis. Geneva: WHO.